Tramadol Infusion 07FEB2019

Protocol AVE-901-104 Phase 3 Open-Label Avenue Therapeutics, Inc.



### STATISTICAL ANALYSIS PLAN

### A PHASE 3, MULTICENTER, SINGLE-ARM, OPEN-LABEL STUDY TO EVALUATE THE SAFETY OF TRAMADOL INFUSION (AVE-901) IN THE MANAGEMENT OF POSTOPERATIVE PAIN FOLLOWING SURGERY PROTOCOL AVE-901-104

Protocol Version 1.0 (11DEC2017)

### SPONSORED BY

Avenue Therapeutics, Inc. New York, NY 10014

### PREPARED BY

Lotus Clinical Research®, LLC 100 W California Blvd, Unit 25 Pasadena, CA 91105 626-397-2390 office info@LotusCR.com www.LotusCR.com

This document is confidential and proprietary to **Avenue Therapeutics**, **Inc.** Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein will be reproduced, published, or otherwise disclosed without the prior written approval of **Avenue Therapeutics**, **Inc.**, except that this document may be disclosed to appropriate Institutional Review Boards under the condition that they keep the information confidential.

Tramadol Infusion 07FEB2019

Protocol AVE-901-104 Phase 3 Open-Label Avenue Therapeutics, Inc.

### **DOCUMENT VERSION CONTROL**

| Version Number | Date | Comments/Changes |
|---|---|---|
| v0.1 | 07SEP2018 For Statistical Review | |
| v0.2 | 12OCT2018 | Update per sponsor feedback |
| v0.3 | 12DEC2018 | Update per sponsor feedback |
| v1.0 | 07FEB2019 | Update per sponsor feedback |

Tramadol Infusion 07FEB2019

### **APPROVALS**

| Author: | DocuSigned by: Sowy Liou Signer Name: Song Liou Signing Reason: I am the author of this document Signing Time: 2/8/2019 2:23:37 PM PST 85C80776CFA1404FB9C34B43BB0AA100 | 08-Feb-19 |
|---|---|---|
| | Song Liou<br>Biostatistician<br>Lotus Clinical Research®, LLC | Date |
| Reviewed: | DocuSigned by: Jennifer Neyer | 08-Feb-19 |
| | Jennifer Nezzer Director, Biometrics Lotus Clinical Research®, LLC | Date |
| Approved: | DocuSigned by: Mike Kyan Signer Name: Mike Ryan Signing Reason: I approve this document Signing Time: 2/11/2019 11:58:34 AM PST 98E11534E6654F4CB5631912227540F0 | 11-Feb-19 |
| | Michael Ryan Vice President Avenue Therapeutics, Inc. | Date |

Tramadol Infusion 07FEB2019

### **APPROVALS**

| Approved: (cont.) | DocuSigned by: Scalt Kinus, MD Signer Name: Scott Reines, MD Signing Reason: I approve this document Signing Time: 2/11/2019 5:36:33 PM PST A89AE03A57484F3F94C5585073F8D59F | 11-Feb-19 |
|---|---|---|
| | Scott Reines Chief Medical Officer Avenue Therapeutics, Inc DocuSigned by: | Date |
| | Signer Name: Lucy Lu, MD Signing Reason: I approve this document Signing Time: 2/11/2019 6:48:28 PM PST 5DDA3F62E50E4ABBBCEE9D8284AEA67B | 11-Feb-19 |
| | Lucy Lu Chief Executive Officer Avenue Therapeutics, Inc. | Date |
| | DocuSigned by: Mark: Harwitt Signer Name: Mark Harnett Signing Reason: I approve this document Signing Time: 2/12/2019 4:19:58 AM PST 0D9F4DA52C0A4BDD8A63BE5F1FE45B64 | 12-Feb-19 |
| | Mark Harnett Tramadol Program Biostatistician Avenue Therapeutics, Inc. | Date |

### **TABLE OF CONTENTS**

| LIST OF | F ABBREVIATIONS | 8 |
|---------|------------------------------------------------|----|
| 1. | PURPOSE OF THE ANALYSES | 9 |
| 2. | PROTOCOL SUMMARY | 10 |
| 2.1. | Study Objectives | 10 |
| 2.1.1. | Primary Objective | 10 |
| 2.2. | Overall Study Design and Plan | 10 |
| 2.3. | Description of Study Periods | 10 |
| 2.3.1. | Screening | 11 |
| 2.3.2. | Preoperative | 11 |
| 2.3.3. | Surgery | 11 |
| 2.3.4. | Treatment Period/ Post Surgery | 11 |
| 2.3.5. | Follow up: | 12 |
| 2.4. | Study Population | 12 |
| 2.5. | Treatment Regimens | 12 |
| 2.5.1. | Study Material | 12 |
| 2.5.2. | Comparator Group | 12 |
| 2.6. | Treatment Assignment and Randomization | 13 |
| 2.7. | Sample Size Determination | 13 |
| 3. | GENERAL ANALYSIS AND REPORTING CONVENTIONS | 14 |
| 4. | PATIENT SUMMARIES | 16 |
| 4.1. | Analysis Populations | 16 |
| 4.2. | Disposition of Patients | 16 |
| 4.3. | Protocol Deviations | 16 |
| 5. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 18 |
| 5.1. | Demographics and Baseline Characteristics | 18 |
| 5.2. | Medical History | 18 |
| 5.3. | Prior and Concomitant Medications | 18 |
| 6. | MEASUREMENTS OF TREATMENT EXPOSURE | 20 |

## Tramadol Infusion 07FEB2019

| 7. | OVERVIEW OF ANALYSIS ISSUES | 21 |
|---------|-----------------------------------------------------|----|
| 7.1. | Handling of Dropouts or Missing Data | 21 |
| 7.2. | Assessment Time Windows | 21 |
| 8. | EFFICACY EVALUATION | 22 |
| 8.1. | Efficacy Outcome | 22 |
| 9. | SAFETY EVALUATION | 23 |
| 9.1. | Overview of Safety Analysis Methods | 23 |
| 9.2. | Adverse Events | 23 |
| 9.2.1. | Subgroups | 27 |
| 9.3. | Deaths and Serious Adverse Events | 27 |
| 9.4. | Clinical Laboratory Evaluation | 27 |
| 9.5. | Vital Signs | 29 |
| 9.6. | Physical Examination | 30 |
| 9.7. | ECG Examinations | 30 |
| 10. | PHARMACOKINETIC EVALUATION | 32 |
| 11. | INTERIM ANALYSES AND DATA MONITORING | 33 |
| 12. | CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL | 34 |
| 13. | REFERENCES | 35 |
| 14. | APPENDICES | 36 |
| 14.1. | Tables, Figures and Listings for Final Study Report | 36 |
| 14.1.1. | Tables | 37 |
| 14.1.2. | Figures | 41 |
| 14.1.3. | Listings | 42 |
| 15. | DOCUMENT HISTORY | 43 |

Tramadol Infusion 07FEB2019

Protocol AVE-901-104 Phase 3 Open-Label Avenue Therapeutics, Inc.

### LIST OF TABLES

| Table 1: | Protocol-Specified Visits and Visit Windows (Study AVE-901-104) | 12 |
|---|---|---|
| Table 2: | Table of Imputation Rules for Missing AE Start Date Times (Study AVE-901-104) | 26 |
| Table 3: | List of Potentially Clinically Significant Ranges for Clinical Laboratory Parameters (Study AVE-901-104) | 28 |
| Table 4: | List of Potentially Clinically Significant Ranges for Vital Sign Parameters (Study AVE-901-104) | 29 |
| Table 5: | List of Potentially Clinically Significant Ranges for ECG Parameters (Study AVE-901-104) | 30 |

### LIST OF ABBREVIATIONS

| ADaM | Analysis Data Model |
|--------|----------------------------------------------|
| AE | Adverse Event |
| ALT | Alanine aminotransferase |
| ASA | American Society of Anesthesiologists |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| CDER | Center for Drug Evaluation and Research |
| eCRF | Electronic Case Report Form |
| CSR | Clinical Study Report |
| ECG | Electrocardiogram |
| EOT | End of Treatment |
| FDA | Food and Drug Administration |
| ICH | International Conference on Harmonization |
| IV | Intravenous |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PCS | Potential Clinically Significant |
| PE | Physical Exam |
| PGA | Patient Global Assessment |
| PT | Preferred Term |
| SAE | Serious Adverse Event/Experience |
| SAP | Statistical Analysis Plan |
| SDTM | Standard Data Table Model |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |

Tramadol Infusion 07FEB2019

### 1. PURPOSE OF THE ANALYSES

This statistical analysis plan (SAP) is based on protocol number AVE-901-104 Amendment 1.0 (29AUG2018) from Avenue Therapeutics, Inc. The SAP will be signed off before the final database lock. The SAP contains detailed information to aid in the performance of the statistical analysis and reporting of the study data for use in the final clinical study report (CSR). This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonization (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials, the most recent ICH E3 Guideline and the Guidance for Industry: Structure and Content of Clinical Study and the most recent FDA draft Guidance for Industry - Analgesic Indications: Developing Drug and Biological Products, dated February 2014.

This SAP describes the data sets that will be analyzed and the patient characteristics, safety, and efficacy assessments that will be evaluated. This SAP provides details of the specific statistical methods that will be used. If additional analyses are performed after database lock to supplement the planned analyses described in this SAP, they will be completed and will be clearly identified as post-hoc in the CSR.

Tramadol Infusion 07FEB2019

Protocol AVE-901-104 Phase 3 Open-Label Avenue Therapeutics, Inc.

### 2. PROTOCOL SUMMARY

### 2.1. Study Objectives

### 2.1.1. Primary Objective

The primary objective of this study is to evaluate the safety of intravenous (IV) tramadol (AVE-901) 50 mg for the management of postoperative pain.

Safety endpoints will include

- Adverse event (classified by the Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC) and preferred term (PT)).
- Clinical laboratory, vital sign, and electrocardiogram (ECG) changes.
- Local tolerability of the infusion site via pain, swelling, tenderness, and erythema.

### 2.2. Overall Study Design and Plan

This study is a Phase 3, multicenter, single-arm, open-label, repeat-dose trial to assess the safety of AVE-901 in the management of postoperative pain. Eligible patients will be patients that are undergoing elective surgery and are willing to be confined in a healthcare facility and receive AVE-901 for the treatment of post-surgical pain for at least 24 hours. Approximately 250 patients will be enrolled into the study. Each patient will undergo the Screening Visit (Day -28 to Day -1), the Pre-operative assessment (within 24 hours prior to surgery), the Surgery (Day 0), the Primary treatment period (hour 0 through hour 168), end of treatment (EOT) visit, and the Follow-up Visit (Day 14).

Screening will occur up to 28 days prior to surgery. Following the pre-operative assessments, after the patient has met eligibility criteria, patients will be enrolled into the study.

Surgery will occur on Day 0. There are no restrictions on the agents to be used for induction, neuromuscular blockade, maintenance of anesthesia, or on hypnotics, sedatives, analgesics (including narcotics) or anxiolytics.

Following surgery, each patient will receive their study medication infusion at T0, T2, T4, and then every 4 hours for up to 168 hours after the first study drug administration (a total of up to 43 doses per patient). The dosing time point will always be defined relative to T0 for all doses. The latest (last) dose that is allowed is at Hour 164. Patients will be confined at an appropriate healthcare or research facility for as long as they are still using AVE-901. Following the first dose of study drug, the patients will be allowed to use non-opioid-based analgesics per treating physician's discretion, if additional pain relief is required.

### 2.3. Description of Study Periods

There are 5 periods in this study: Screening, Preoperative, Surgery, Treatment Period/Post Surgery, and Follow-up. Procedures for each study period are described below.

Tramadol Infusion 07FEB2019

### 2.3.1. Screening

Screening will occur from Day -28 through Day -1 and will be conducted as a clinic visit. Patients will have the purpose and procedures of the study explained to them and, those who elect to participate in the study, will provide written informed consent and be screened for participation according to the eligibility criteria. Screening will include eligibility assessment, medical history, physical examination (PE), demographics, height and weight, body mass index (BMI), vital signs (heart rate, systolic blood pressure (BP), and diastolic BP, respiratory rate, temperature, pulse oximetry), American Society of Anesthesiologists (ASA) Physical Status, 12lead ECG, hematology panel, chemistry panel, urinalysis, serum pregnancy test (in females of childbearing potential), and prior/current treatments. All screening laboratory evaluations must be within acceptable limits as determined by the investigator prior to enrollment. For patients that screen within 5 days of surgery, central laboratory values may not be available to assess eligibility. For these patients it is acceptable for sites to draw local labs to assess eligibility in addition to the central lab which will still be used as the baseline in the study. The local laboratory listed on the FDA 1572 Form must be used for all local blood draws. At a minimum the following analytes must be reviewed from the local laboratory prior to dosing; magnesium, calcium, potassium, sodium, serum creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST) and hemoglobin.

### 2.3.2. Preoperative

Preoperative assessments to confirm the patient's eligibility will be performed within 24 hours of scheduled surgery start time. This visit will include reassessment of eligibility criteria, interim medical history, vital signs, PE, ASA Physical Status, urine pregnancy test (in females of childbearing potential), and concomitant treatments.

Note: If the patient's scheduled surgery has time considerations, patients may have Screening and Preoperative Visits combined into one visit if required (at the time of pre-op). The procedures associated with the Screening Visit will be acceptable for both visits. Both central and local labs should be drawn for eligibility

### 2.3.3. Surgery

Surgery will occur on Day 0. Sites will follow their standard operating procedures.

### 2.3.4. Treatment Period/ Post Surgery

Patients will receive their first dose of study medication (T0) within 8 hours of meeting the postsurgical eligibility criteria. Patients will be dosed at Hour T0, T2, T4, and then every 4 hours thereafter, for a total of up to 43 doses administered over the 168-hour treatment period (with the last possible dose at Hour 164). Treatment is anticipated to occur from Hours 0 to 48 and may extend through to Hour 168.

Safety will be assessed by recording vital signs including: ECG's, respiratory rate, heart rate, pulse oximetry (SpO2), temperature, and BP as per the schedule of events.

A PGA will be obtained at Hour 24 and EOT. If the patient continues treatment beyond Hour 24, CONFIDENTIAL

Tramadol Infusion 07FEB2019

PGA will be conducted at Hour 24 and EOT (total of 2 PGAs). If the patient ends treatment prior to Hour 24, PGA will be conducted as part of the EOT visit (total of 1 PGA).

At the EOT assessment, patients will undergo a brief PE, vital signs measurements, ECG, PGA and clinical laboratory evaluations for safety. AEs and concomitant medication use will be recorded.

### **2.3.5.** Follow up:

A final safety assessment will be conducted on Day 14 ( $\pm$  2 days) from the first dose via a telephone call to check on general well-being, including spontaneous reports of adverse events and concomitant medications.

The protocol-defined visits are presented in Table 1.

Table 1: Protocol-Specified Visits and Visit Windows (Study AVE-901-104)

| Study Phase | Visit Time |
|---|---|
| Screening | From days -28 to -1 |
| Pre-Operative | 0 - 24 Hours prior to surgery |
| Surgery | Day 0 |
| Treatment Period /Post Surgery | Hours 0 up to Hour 168 after infusion of first study drug administration |
| Follow-up | Day 14 (approximately Day 14±2 days) |

### 2.4. Study Population

Approximately 250 patients in United States (US) who meet all the inclusion and none of the exclusion criteria (Described in Sections 7.1, 7.2 and 7.2.1 of Protocol) are planned to be enrolled. Every patient treated will receive AVE-901.

### 2.5. Treatment Regimens

### 2.5.1. Study Material

AVE-901, 50 mg. Assigned study treatment (51 mL) doses will be administered IV over 15 minutes (+/- 4 minutes) via infusion pump.

All patients will receive tramadol infusion per the treatment dosing regimen. A trained health care professional will flush the line with normal saline at the end of each infusion. Throughout the SAP, AVE-901 will be used to indicate the study treatment.

### 2.5.2. Comparator Group

NA as this is a single arm study.

Tramadol Infusion 07FEB2019

### 2.6. Treatment Assignment and Randomization

No randomization will be utilized in this study.

### 2.7. Sample Size Determination

A sample size of approximately 250 patients will be enrolled. This sample size of 250 patients will provide approximately 90% power to detect at least one incidence of uncommon adverse events (those events with a true underlying incidence of 1%).

Tramadol Infusion 07FEB2019

### 3. GENERAL ANALYSIS AND REPORTING CONVENTIONS

This section discusses general policies to be employed in the analysis and reporting of the data from the study. Departures from these general policies are provided in the specific detailed sections of this SAP. When this situation occurs, the rules set forth in the specific section take precedence over the general policies.

All continuous study assessments will be summarized by time point (as applicable) using the descriptive statistics n, mean, SD, median, and range (minimum, and maximum). All of the categorical study assessments will be summarized by time point (as applicable) using frequency counts and rates of occurrence (%).

The treatment group will be labeled as 'Tramadol 50 mg' for all outputs. All study data will be listed by study center, patient, and time point (as applicable).

No preliminary rounding will be performed; rounding will only occur after the analysis. To round, consider the digit to the right of the last significant digit: if <5, then round down; if  $\ge 5$ , then round up. Means and medians will be presented with one more decimal place than the precision of the raw data. Standard deviations will be presented with two more decimal places than the precision of the raw data. Percentages will be presented with one decimal place. Minimums and maximums will be presented with the same precision as the original data.

All analyses will be performed using the SAS System® version 9.3 or higher. The domain (Study data tabulation Model [SDTM]) and analysis (Analysis Data Model [ADaM]) data sets will be taken as input to the SAS programs that generate the report-ready tables, figures and listings. The submission ready SDTM and ADaM data sets will be provided to the sponsor along with display deliveries.

The following conventions will be used throughout the study analysis:

- Time T0 is the time of start of the first study drug administration.
- Study Day is defined as (Date of Assessment minus Date of First Dose of Study Medication). The first day of dosing is Study Day 0. The day immediately prior to first dose is Study Day -1. Study Day will be calculated for every record in the database and presented alongside the date fields in the data listings, where applicable. For instance, the start *date* of each TEAE will also have the Start *Day* presented in the listings.
- Assessment and visit times are defined relative to time T0.
- Baseline value is defined as the last valid measurement prior to the first treatment administration.
- Change from baseline is defined as post-baseline value minus baseline value.
- Unscheduled visits and measurements will be included in subject listings but will not be used in analyses.

Tramadol Infusion 07FEB2019

- If duplicate values are obtained at a given visit (e.g., lab assay is repeated on a sample resulting in two results, or vital sign repeated during a visit), the last reported value will be used unless it is noted that the measurement was in error for that value.
- Values that compromise interpretation will not be used in summaries (e.g., values that were obtained post-dose will not be summarized as pre-dose values).

Tramadol Infusion 07FEB2019

Protocol AVE-901-104 Phase 3 Open-Label Avenue Therapeutics, Inc.

### 4. PATIENT SUMMARIES

### 4.1. Analysis Populations

Three population are identified for purposes of the statistical analysis:

- Screened Population, defined as all screened patients.
- Screened Not Treated, defined as the subset of patients who are screened but not treated due to not moving forward to surgery or not meeting post-surgical dosing criteria.
- The Safety Population is defined as all patients who receive study medication. Patients will be analyzed according to the actual treatment they receive.

In general, data listings will include only subjects who receive study treatment (Safety population).

### 4.2. Disposition of Patients

Disposition of all patients screened will be tabulated. The Inclusion/Exclusion criteria failed for screen failures will be presented. The denominator will be based on all screened patients.

Patient completion status (completer, screen failure, or post-op failure) and reasons for study completion will be tabulated descriptively in a patient disposition summary table. Reasons for study completion include:

- Dosing Completed (patient discharged and did not stop dosing for the other items listed below)
- Adverse Event
- Lost to Follow-Up
- Death
- Protocol Violation
- Subject Non-compliance or uncooperativeness
- Withdrawal of Consent
- Other

The number of days in the study will also be summarized. The number of days is computed as: [Date of study completion (i.e., date of discharge) or withdrawal minus the date of first treatment administration (Day 1)] + 1.

All patient disposition data will be presented in listings.

### 4.3. Protocol Deviations

Protocol deviations will be documented in the electronic case report from (eCRF), categorized according to type of deviation (e.g., out of window, etc.) and classified as major or minor by the Sponsor's medical monitor. Protocol deviations, both minor and major, will be presented in a

Tramadol Infusion 07FEB2019

data listing and major violations will be summarized by category of deviation and classification. A listing describing patients excluded from the Per Protocol Population will be provided.

Tramadol Infusion 07FEB2019

### 5. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

### **5.1.** Demographics and Baseline Characteristics

Demographic variables include age, sex, race, and ethnicity. Baseline characteristics include American Society of Anesthesiologists (ASA) physical status, previous opioid history (Y/N), height, weight (kg) and BMI (kg/m²). Demographics and baseline characteristics will be presented in by-patient listings and summarized.

### **5.2.** Medical History

Medical history, as collected at screening and prior to surgery, will be presented in a by-patient listing and summarized by body system.

### **5.3.** Prior and Concomitant Medications

Prior and concomitant medications are collected at screening and updated throughout the study as needed. Prior and concomitant medications will be coded using WHODDE (C Format) version 01SEP2017. The number and percentage of patients who take concomitant medications will be summarized by drug class (Anatomical Therapeutic Chemical (ATC) Level 3) and PT for the safety population and presented in a by-patient listing.

Prior medications, including medications given during surgery, and non-medical therapies will appear in a data listing but will not be summarized.

Medications will be classified as follows:

- Prior medications. Prior medications/therapies are those that have a start date/time and end date/time prior to the start of the first treatment administration. Prior medications will not be tabulated but will be included in the data listings.
- Concomitant medications. Medications will be considered as concomitant if the medication is taken on or after the date/time of first intake of treatment product and has a start date/time that is no later than 1 day (24 hours) after the start of the last administration of study medication.
- New-onset concomitant medications are defined as those medications starting between the start of the first dose of study medication and 1 day (24 hours) after the start of the last dose of study medication. Medications with no start time but starting on the day of study medication will be assumed to be new-onset.
- Post-treatment medications. Post-treatment medications are defined as a medication with a start date/time at least 24 hours (1 day) after the start of the last dose of study medication.

If a missing medication start date cannot be definitively determined as having started after first dose, the medication will be considered as started prior to first dose; similarly, if a missing medication stop date/time cannot be determined as having stopped prior to first dose, the medication will be considered concomitant (taken after first dose). Imputation of missing start CONFIDENTIAL

Tramadol Infusion 07FEB2019

and stop date/times will be performed in the same manner as described for AEs in Table 2. Medications with entirely missing start and stop dates will be listed but not included in the tabulations.

Tramadol Infusion 07FEB2019

### 6. MEASUREMENTS OF TREATMENT EXPOSURE

Patient dosing data will be listed and the number of doses per subject and total exposure (mg) per subject will be tabulated. If less than the complete volume of study medication is infused, total exposure will be calculated as the intended dosage (50mg) times the proportion of total saline volume infused (xx mL / 50 mL).

- The duration of exposure will be defined in hours, in which the time from the start of the first dose to start of the last dose, plus 4 hours (i.e., exposure is assumed to be 4 hours for each dose), will be tabulated.
- The number (%) of patients by number of doses received will be presented. The maximum total number of doses is 43.
- The total exposure (mg) will be summarized through 24, 48, 72, 96, 120, 144 and 164 hours, respectively. Maximum exposure is 2150 mg (given at Hours 0, 2, 4, and then 4 hours up to 164).
- If infusion end time is not available, the end time will be imputed as 15 minutes after the infusion start time for use in calculations dependent upon the end time.

In addition, cumulative percent of subjects (%) versus total study drug exposure will be provided graphically.

Tramadol Infusion 07FEB2019

### 7. OVERVIEW OF ANALYSIS ISSUES

No inferential testing is planned for this safety-based single arm study.

### 7.1. Handling of Dropouts or Missing Data

No study outcomes will be imputed.

### 7.2. Assessment Time Windows

Summaries will be based on the nominal protocol-specified visits as appropriate.

Tramadol Infusion 07FEB2019

### 8. EFFICACY EVALUATION

The primary objective of this study is to evaluate the safety of AVE-901. Efficacy is considered a secondary, exploratory, given that this is an uncontrolled study in patients with various surgery types. Efficacy will be assessed by patient global assessments (PGAs) using a 5-point scale.

### 8.1. Efficacy Outcome

Patient Global Assessment of efficacy will be collected at 24 hours post first dose and EOT. The question to be posed is "How would you rate the study medication in terms of its effectiveness in controlling your pain?" (0=poor; 1=fair; 2=good; 3=very good; 4=excellent). If the patient continues treatment beyond Hour 24, PGA will be conducted at Hour 24 and EOT (total of 2 PGAs). If the patient ends treatment prior to Hour 24, PGA will be conducted as part of the EOT visit (total of 1 PGA).

The PGA results will be presented in a summary table by time point. The number (%) of subjects answering in each category will also be presented by time point.

Individual PGA scores will be listed

### 9. SAFETY EVALUATION

### 9.1. Overview of Safety Analysis Methods

The safety analysis will be descriptive in nature. All safety data will be listed, and data will be tabulated where the data warrant. Safety data include:

- AEs, including assessment of infusion site local reactions (skin and vein)
- Clinical laboratory tests (hematology panel, chemistry panel and urinalysis) pretreatment and discharge
- Vital signs including: respiratory rate, heart rate, oral temperature, pulse oximetry (SpO2) and BP, as per the schedule of events
- PE at pre-treatment and discharge
- 12-lead ECG at protocol specified time points
- Concomitant treatments

Anti-emetic usage data will be included with the concomitant treatments. Exploratory analyses of use of anti-emetics may be performed if warranted. Other safety data presentations will be descriptive in nature and no formal statistical tests will be performed.

ECG results will be analyzed on an ongoing basis by a central ECG reader on an individual patient level.

### 9.2. Adverse Events

Any events starting before the first dose of treatment will be reported as Medical History. Verbatim terms used by investigators to identify AEs in the CRFs will be mapped to the appropriate PT and SOC using a standardized coding dictionary (MedDRA Version 20.1). All coding will be reviewed prior to database lock. All recorded AEs will be listed; adverse events starting on or after the first dose of treatment are considered treatment-emergent adverse events as per the protocol, but the definition of treatment emergent will be further categorized for summaries as follows:

- Adverse events occurring on or after the first dose of study medication, and within 1 day (up to 24 hours) after the start of the last dose of study medication. For simplicity, these will be referred to as Treatment Emergent AEs (TEAEs) in the summaries.
- Events occurring after that will be presented as Post-Treatment AEs.

Separate tabulations will be presented for TEAEs and for Post-Treatment AEs.

For evaluation of causal relatedness to treatment, the categories are definite, probable, possible, remote or definitely not. For categorization in the summary tables, AEs designated as definite, probable, or possible will be considered to be related.

For the evaluation of event severity, the criteria are based on National Cancer Institute Common

Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03:

| CTC Grade | CTCAE Grade Description |
|---|---|
| Grade 1: Mild | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |
| | observations only; intervention not indicated. |
| Grade 2: Moderate | Minimal, local or noninvasive intervention indicated; limiting age- |
| | appropriate instrumental ADL <sup>1</sup> . |
| Grade 3: Severe | Severe or medically significant but not immediately life- |
| | threatening; hospitalization or prolongation of hospitalization |
| | indicated; disabling; limiting self-care ADL <sup>2</sup> . |
| Grade 4: Life-threatening | Life-threatening consequences; urgent intervention indicated. |
| Grade 5: Death | Death related to the AE. |

<sup>&</sup>lt;sup>1</sup> ADL = Activities of Daily Living. Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

Local tolerability at the infusion site will be assessed for pain, swelling, tenderness, and erythema. Any such AEs related to tolerability at the infusion site will be identified by the sponsor and medical monitor for listing and possible summarization.

In addition to a listing of all TEAEs, treatment related TEAEs, serious TEAEs, TEAEs leading to premature discontinuation from the study, and TEAEs related to local tolerability at the infusion site will be provided.

An overall summary will be prepared including both the number of TEAEs, and the number of patients with TEAEs, as well as SAEs, treatment related TEAEs, TEAEs by severity and TEAEs leading to premature discontinuation from study.

Incidence of TEAEs will be summarized by SOC and PT sorted in descending frequency by SOC, and then by PT within SOC. These summaries will be given in separate tables for each of the following TEAE event sets:

- All events (Post-Treatment AEs will be tabulated separately)
- Treatment related events (defined by a relationship to study drug of possible, probable, or definite). (Post-Treatment AEs will be tabulated separately)
- Events leading to premature discontinuation from study
- Events related to local tolerability at the infusion site
- Events by maximum severity

If a given patient experiences a TEAE that maps to the same PT more than once, the patient will be counted once for the PT at its greatest severity (i.e., mild, moderate, or severe) and causality

<sup>&</sup>lt;sup>2</sup> Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

Tramadol Infusion 07FEB2019

(i.e., attribution to study material).

TEAEs occurring within 1 hour of any infusion will be summarized.

The number/ percentages of subjects with any TEAE will also be presented by Infusion #. Each AE will be matched to an Infusion # by the start date/time of the AE (after all imputation for missing dates). E.g., An AE with start date/time on or after the start date/time of Infusion #3 and prior to start date/time of Infusion #4, will be counted under Infusion #3. Percentages will be calculated from the number of subjects receiving the referenced injection (i.e., Subjects receiving 4 injections will be counted in the denominator for Infusion #1, #2, #3 and #4, and will not be included in the denominator for other Infusions).

Duration of a TEAE will be computed in days as the stop date of the event minus the start date plus 1. If reported as ongoing at the time of database lock, the duration of the AE will be calculated using the date/time of the last visit or the last date of any adverse event for the patient in the database, whichever is later. If a TEAE is considered resolved, but the stop date is missing, the last day of the month will be imputed if the month and year are available. If only the year is available, and the year is the same as the year of the last visit, the stop date will be imputed as the latest of the last visit date or latest event for the patient in the database. If the year of the event is prior to the year of the last treatment, the end day and month will be imputed as 31 December.

For missing or partial start dates, they will be imputed as temporally related to the first dose of study medication. Table 2 demonstrates the rules to be used to impute any missing AE start dates.

Table 2: Table of Imputation Rules for Missing AE Start Date Times (Study AVE-901-104)

| Missing Start Date<br>Portion | Prior to<br>Treatment | Same as<br>Treatment Start<br>Date | After Treatment Start<br>Date |
|---|---|---|---|
| Day | Month and Year < Month and Year of first treatment: | Month and Year = Month and Year of first treatment: | Month and Year ><br>Month and Year of<br>First Treatment: |
| | Start Day = 1 | Start Day = Day of | Start Day = 1 |
| | Stop Day = last day of the month | first treatment Stop Day= last day of the month | Stop Day= last day of the month |
| Day and Month<br>Define Day as<br>above, then: | Year < Year of first treatment: | Year = Year of first treatment: | Year > Year of first treatment: |
| | Start Month = July | Start Month = | Month = January |
| | Stop Month = Dec | Month of first treatment | Stop Month = Dec |
| | | Stop Month = $Dec$ | |
| Day, Month, and<br>Year | To be conservative, completely missing start dates will be set to the date of first treatment, completely missing end dates will be set to the date of last contact. | | |
| Time | Missing start times will be imputed as 00:01 (or the start time of the first dose administration if AE occurred on the date of first dose administration) | | |
| | Missing stop times will b | e imputed as 23:59 | |

After following these imputation rules, if the start date/time is imputed as a date after the end date/time, the start date/time will be set to the end date/time to provide a positive duration for the event incidence.

Missing assessments for AE study medication relationship or severity will be analyzed as related or severe respectively. No other imputation is planned for safety data.

Tramadol Infusion 07FEB2019

### 9.2.1. Subgroups

Descriptive analysis of treatment-emergent AEs (TEAEs), serious adverse events (SAEs), and discontinuations due to AEs, will be provided by the following subgroups:

- Gender (male versus female)
- Race (White versus non-White)
- Age (using the study median age: less or equal to (≤) median age group versus greater than (>) median age group)
- Age (<65 vs>=65 years)
- BMI (> versus <= median value)
- Surgery Type (Orthopedic versus soft tissue)

### 9.3. Deaths and Serious Adverse Events

A serious adverse event is an AE occurring during the study that fulfills one or more of the following:

- Results in death
- It is immediately life-threatening
- It requires in-patient hospitalization or prolongation of existing hospitalization
- It results in persistent or significant disability or incapacity
- Results in a congenital abnormality or birth defect
- It is an important medical event that may jeopardize the patient or may require medical intervention to prevent one of the outcomes listed above

Serious adverse events and deaths will be listed and summarized separately for the safety population.

### 9.4. Clinical Laboratory Evaluation

Clinical laboratory test results (blood chemistry, hematology and urinalysis) will be listed for individual patients. Baseline for clinical laboratory parameters will be defined as the last evaluation before dosing with study treatment. For each individual lab test value, results and change from baseline will be summarized by time point (baseline and at discharge).

The number and percent of patients with potentially clinically significant (PCS) values will be summarized. Only new-onset PCS values, i.e., patients with pre-existing PCS values at pre-treatment will not be considered to have new-onset values on-treatment. The criteria used to identify potentially clinically significant laboratory values are listed in Table 3.

Table 3: List of Potentially Clinically Significant Ranges for Clinical Laboratory Parameters (Study AVE-901-104)

| Variable Name (Normal Range) | Low | High |
|---|---|---|
| Hematology | | |
| White Blood Cells (NR: 3.7 - 11.0x K/cu/mm) | $\leq 2.8 \text{ x } 10^3 \text{ /mm}^3$ | $\geq 16 \times 10^3 / \text{mm}^3$ |
| Neutrophils (NR: 46 - 72%) | ≤ 15% | NA |
| Lymphocytes (NR: 14 - 46%) | NA | ≥75% |
| Monocytes (NR: 0 - 11%) | NA | ≥15% |
| Eosinophils (NR: 0 - 7%) | NA | ≥10% |
| Basophils (NR: 0 - 3%) | NA | ≥10% |
| Red Blood Cells<br>Female: (NR: 3.8 - 5.1 x 10 <sup>6</sup> /mm <sup>3</sup> )<br>Male: (NR: 4.1 - 5.6 x 10 <sup>6</sup> /mm <sup>3</sup> ) | ≤3 x 10 <sup>6</sup> /mm <sup>3</sup><br>≤3.5 x 10 <sup>6</sup> /mm <sup>3</sup> | $\geq$ 6 x 10 <sup>6</sup> /mm <sup>3</sup> $\geq$ 6.5 x 10 <sup>6</sup> /mm <sup>3</sup> |
| Hematocrit | | |
| Female: (NR: 36.4 – 48.9%) | ≤32% | NA |
| Male: (NR: 41.6 – 54.1%) | ≤37% | NA |
| Hemoglobin | | |
| Female: (NR: 11.5 – 16.0 g/dL) | ≤9.5 g/dL | NA |
| Male: $(NR: 13.0 - 17.5 \text{ g/dL})$ | $\leq 11.5 \text{ g/dL}$ | NA |
| Platelets (NR: 125 - 375 K/cu/mm) | $\leq 75 \text{ x } 10^3 \text{ /mm}^3$ | $\geq$ 700 x 10 <sup>3</sup> /mm <sup>3</sup> |
| Serum Chemistry | | |
| Total protein (NR: 6.0 - 8.0 g/dL) | ≤4.0 g/dL | ≥10 g/dL |
| Albumin (NR: 3.5 - 5.5 g/dL) | $\leq 2.0 \text{ g/dL}$ | NA |
| Creatinine (NR: 0.7 - 1.4 mg/dL) | NA | ≥2 mg/dL |
| BUN (NR: 5 - 20 mg/dL) | NA | ≥30 mg/dL |
| Uric Acid: (NR: 2.0 - 6.0 mg/dL | NA | $\geq$ 9.0 mg/dL |
| Bilirubin total (NR: 0.1 – 1.1 mg/dL) | NA | ≥2.5 mg/dL |
| Bilirubin direct (NR: 0 - 0.4 mg/dL) | NA | $\geq$ 0.6 mg/dL |
| Alkaline phosphatase (NR: 30 - 115 U/L) | NA | ≥390 IU/L |
| AST/SGOT | NA | □150 U/L |
| ALT/SGPT | NA | □165 U/L |
| CPK (NR: 24 - 169 U/L) | NA | ≥702 IU/L |
| Glucose random (NR: 60 - 115 mg/dL) | ≤40 mg/dL | ≥250 mg/dL |
| ` | | |

| Variable Name (Normal Range) | Low | High |
|---|---|---|
| Phosphorous (NR: 2.5 - 4.5 mg/dL) | ≤1.7 mg/dL | NA |
| Sodium (NR: 133 - 145 mEq/L) | $\leq$ 126 mEq/L | ≥156 mEq/L |
| Potassium (NR: 3.5 - 5.0 mEq/L) | ≤3 mEq/ | ≥6 mEq/L |
| Chloride (NR: 95 - 110 mEq/L) | ≤90 mEq/L | ≥118 mEq/L |
| Bicarbonate (CO <sub>2</sub> ) (NR: 21 - 33 mEq/L) | ≤19 mEq/L | ≥35 mEq/L |
| Urinalysis | | |
| Specific gravity (NR: 1.002 - 1.035) | ≤1.001 | NA |
| pH (NR: 5.0 – 8.0) | ≤4 | ≥9 |
| UA Ketones (Normal = negative) mg/dL | NA | ≥2+ |
| UA Protein (Normal = negative) mg/dL | NA | ≥2+ |
| UA Blood (Normal = negative) | NA | ≥3+ |
| UA Leukocyte Esterase | NA | ≥3+ |
| Nitrates | NA | ≥2 |

Each clinical laboratory test will be defined to be "Low", "Normal", or "High", according to the normal reference range from the clinical laboratory. The number and percentage of patients who have a shift from within to outside the normal reference range from baseline (and vice versa) to each follow-up visit will be summarized by time point.

### 9.5. Vital Signs

Vital signs results including BP (systolic and diastolic), heart rate, respiration rate, pulse oximetry, and temperature will be listed for individual patients. Baseline for vital signs measurements will be defined as the last evaluation before dosing with study medication. Vital signs and changes from baseline will be summarized by time point.

Vital sign parameter outcomes will be assessed for potential clinical significance; observed values and changes from pre-treatment to on-treatment time points will be tabulated for continuous parameters, as warranted.

The number and percent of patients with potentially clinically significant (PCS) values during the treatment phase will be summarized. A focus will be on new-onset PCS values, i.e., patients with pre-existing PCS values at pre-treatment will not be considered to have new-onset values on-treatment. The criteria for identifying potentially clinically significant vital signs values are provided in Table 4.

Table 4: List of Potentially Clinically Significant Ranges for Vital Sign Parameters (Study AVE-901-104)

| Variable Name | LOW | HIGH |
|---------------|-----|------|
|---------------|-----|------|

| Systolic BP | <86 mm Hg OR a decrease of<br>≥25 mm Hg from baseline | >200 mm Hg OR an increase of ≥25 mm Hg from baseline |
|---|---|---|
| Diastolic BP | <48 mm Hg OR a decrease of<br>≥20 mm Hg from baseline | >110 mm Hg OR an increase of ≥20 mm Hg from baseline |
| Heart rate <sup>1</sup> | 1) <45 bpm OR a decrease of ≥25 bpm from baseline | 1) >105 bpm and increase ≥25 bpm from baseline OR >125 bpm |

<sup>&</sup>lt;sup>1</sup>bpm: beats per minute

### 9.6. Physical Examination

Physical examination results will be listed for individual patients.

### 9.7. ECG Examinations

ECG examination interpretation results and heart rate and interval duration results will be listed for individual patients. Baseline for ECG continuous measurements will be defined as the last evaluation before dosing with study medication. Continuous ECG values and changes from baseline will be summarized by time point. The proportion of subjects with Normal, Abnormal: Not Clinically Significant, and Abnormal: Clinically Significant will be summarized by time point.

The ECG analysis will include a careful review of QTcF values. As part of this review, a summary of the number (percent) of patients with QTcF values in the following ranges will be provided:  $\leq$ 450 msec, >450 to  $\leq$ 480 msec, >480 to  $\leq$ 500 msec, and >500 msec. This will be performed by visit as well as at ANY time during the treatment period (where the highest QTcF value will be used for that assessment).

The incidence of PCS values will be presented, with a focus on new-onset PCS values. The criteria for identifying potentially clinically significant ECG values are provided in Table 5.

Table 5: List of Potentially Clinically Significant Ranges for ECG Parameters (Study AVE-901-104)

| PR Interval |
|-----------------------------------------------------|
| High: >200 msec OR Increase ≥ 20 msec from baseline |
| QRS Interval |
| High: >100 msec OR Increase ≥ 10 msec from baseline |
| QT Interval |
| High: >500 msec OR Increase ≥ 60 msec from baseline |
| QTcF Interval |

Tramadol Infusion 07FEB2019

| High: > 450 msec (Males); >470 msec (Females) OR Increase ≥ 50 msec from baseline |
|---|
| Heart Rate |
| Low: <45 bpm OR a decrease of ≥25 bpm from baseline |
| High: >105 bpm and increase ≥25 bpm from baseline OR >125 bpm |

Tramadol Infusion 07FEB2019

### 10. PHARMACOKINETIC EVALUATION

There are no pharmacokinetic assessments being performed in this study.

Tramadol Infusion 07FEB2019

### 11. INTERIM ANALYSES AND DATA MONITORING

There are no planned interim analyses for this study.

Tramadol Infusion 07FEB2019

### 12. CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL

This SAP analysis is consistent with that described in the study protocol, with clarifications and minor modifications to ensure a robust and scientifically valid analysis.

Tramadol Infusion 07FEB2019

### 13. REFERENCES

US Federal Register. (1998) International Conference on Harmonization; Guidance for Industry: Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration. Federal Register, Vol. 63, No. 179, September 16, 1998, page 49583.

US Federal Register. (1996) International Conference on Harmonization; Guidance for Industry: Structure and Content of Clinical Study Reports. Department of Health and Human Services: Food and Drug Administration. Federal Register Vol. 61, July 17, 1996, page 37320.

Guidance for Industry (2014) Analgesic Indications: Developing Drug and Biological Products - Draft Guidance. Department of Health and Human Services: Food and Drug Administration. Center for Drug Evaluation and Research (CDER) February 2014 Clinical/Medical.

DocuSign Envelope ID: 0709CFD0-5808-479E-B07C-DD202170566C

Protocol AVE-901-104 Phase 3 Open-Label Avenue Therapeutics, Inc.

Tramadol Infusion 07FEB2019

# 14. APPENDICES

# 14.1. Tables, Figures and Listings for Final Study Report


Tramadol Infusion 07FEB2019

# 14.1.1. Tables

| Table Number | Table Title | Analysis Populations | Subgroups | Topline | Unique or |
|---|---|---|---|---|---|
| | | | | | Repeat |
| Table 14.1.1 | Summary of Subject Disposition | All Screened Subjects | | | Unique |
| Table 14.1.2 | Summary of Subjects by Study Center | Safety Population | | | Unique |
| Table 14.1.3 | Summary of Major Protocol Deviations | FAS Population | | | Repeat |
| Table 14.1.4 | Summary of Demographic and Baseline Characteristics | FAS Population | | Yes | Unique |
| Table 14.1.5 | Summary of Medical/ Surgical History by Body System | Safety Population | | | Unique |
| Table 14.1.6.1 | Summary of Concomitant Medications by ATC Class and Preferred Term | Safety Population | | | Unique |
| Table 14.1.6.2 | Summary of New-Onset Concomitant Medications by ATC Class and Preferred Term | Safety Population | | | Repeat |
| Table 14.1.7 | Summary of Study Medication Exposure | Safety Population | | Yes | Unique |
| Table 14.2 | Summary of Patient Global Assessment (PGA) | Safety Population | | | Unique |
| Table 14.3.1 | Overall Incidence of Treatment-Emergent<br>Adverse Events | Safety Population | | Yes | Unique |
| Table 14.3.1.1 | Incidence of Treatment-Emergent Adverse Events and Treatment Related Treatment-Emergent Adverse Events by System Organ Class and | Safety Population | | Yes | Unique |
| Table 14.3.1.1.1 | Incidence of Treatment-Emergent Adverse Events and Treatment Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Surgery Type | Safety Population | Surgery Type | | Unique |
| Table 14.3.1.1.2 | Incidence of Treatment-Emergent Adverse Events and Treatment Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Gender | Safety Population | Gender | | Repeat |
| Table 14.3.1.1.3 | Incidence of Treatment-Emergent Adverse Events<br>and Treatment Related Treatment-Emergent<br>Adverse Events by System Organ Class, Preferred<br>Term and Race | Safety Population | Race | | Repeat |


DocuSign Envelope ID: 0709CFD0-5808-479E-B07C-DD202170566C

Protocol AVE-901-104 Phase 3 Open-Label Avenue Therapeutics, Inc.

Tramadol Infusion 07FEB2019

| Table 14.3.1.1.4.1 | Incidence of Treatment-Emergent Adverse Events and Treatment Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Age Group (Median) | Safety Population | Age (<=, ><br>Median) | Repeat |
|---|---|---|---|---|
| Table 14.3.1.1.4.2 | Incidence of Treatment-Emergent Adverse Events and Treatment Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and Age Group (65 Years Old) | Safety Population | Age (<65, >=<br>65 years old) | Repeat |
| Table 14.3.1.1.5 | Incidence of Treatment-Emergent Adverse Events and Treatment Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term and BMI | Safety Population | BMI | Repeat |
| Table 14.3.1.2 | Incidence of Post-Treatment Adverse Events and<br>Treatment Related Post-Treatment Adverse<br>Events by System Organ Class and Preferred<br>Term | Safety Population | | Repeat |
| Table 14.3.1.3 | Incidence of Treatment-Emergent Adverse Events<br>Leading to Discontinuation from Study by System<br>Organ Class and Preferred Term | Safety Population | | Repeat |
| Table 14.3.1.3.1 | Incidence of Treatment-Emergent Adverse Events<br>Leading to Completion from Study by System<br>Organ Class, Preferred Term and Surgery Type | Safety Population | Surgery Type | Repeat |
| Table 14.3.1.3.2 | Incidence of Treatment-Emergent Adverse Events<br>Leading to Discontinuation from Study by System<br>Organ Class, Preferred Term and Race | Safety Population | Gender | Repeat |
| Table 14.3.1.3.3 | Incidence of Treatment-Emergent Adverse Events<br>Leading to Discontinuation from Study by System<br>Organ Class, Preferred Term and Race | Safety Population | Race | Repeat |
| Table 14.3.1.3.4.1 | Incidence of Treatment-Emergent Adverse Events<br>Leading to Discontinuation from Study by System<br>Organ Class, Preferred Term and Age Group<br>(Median) | Safety Population | Age (<=, ><br>Median) | Repeat |
| Table 14.3.1.3.4.2 | Incidence of Treatment-Emergent Adverse Events<br>Leading to Discontinuation from Study by System<br>Organ Class, Preferred Term and Age Group (65<br>Years Old) | Safety Population | Age (<65, >= 65 years old) | Repeat |


DocuSign Envelope ID: 0709CFD0-5808-479E-B07C-DD202170566C

Protocol AVE-901-104 Phase 3 Open-Label Avenue Therapeutics, Inc.

Tramadol Infusion 07FEB2019

| Repeat | Repeat | Repeat | Unique | Unique | Repeat | Repeat | Repeat | Repeat | Repeat | Repeat | Repeat | Repeat |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Yes | | | | | | |
| BMI | | | | | | | Surgery Type | Gender | Race | Age (<=, ><br>Median) | Age (<65, >= 65 years old) | BMI |
| Safety Population | Safety Population | Safety Population | Safety Population | Safety Population | Safety Population | Safety Population | Safety Population | Safety Population | Safety Population | Safety Population | Safety Population | Safety Population |
| Incidence of Treatment-Emergent Adverse Events<br>Leading to Discontinuation from Study by System<br>Organ Class, Preferred Term and BMI | Incidence of Treatment-Emergent Adverse Events<br>Leading to Death by System Organ Class and<br>Preferred Term | Incidence of Treatment-Emergent Adverse Events<br>Related to Local Tolerability at the Infusion Site<br>by Preferred Term | Incidence of Treatment Adverse Events by<br>System Organ Class, Preferred Term and<br>Maximum Severity | Incidence of Treatment-Emergent Adverse Events<br>and Treatment Related Adverse Events by<br>Infusion Number | Incidence of Treatment Adverse Events and<br>Treatment Related Adverse Events within One<br>Hour of Any Infusion by System Organ Class and<br>Preferred Term | Incidence of Serious Adverse Events by System<br>Organ Class and Preferred Term | Incidence of Serious Adverse Events by System<br>Organ Class, Preferred Term and Surgery Type | Incidence of Serious Adverse Events by System<br>Organ Class, Preferred Term and Gender | Incidence of Serious Adverse Events by System<br>Organ Class, Preferred Term and Race | Incidence of Serious Adverse Events by System<br>Organ Class, Preferred Term and Age Group<br>(Median) | Incidence of Serious Adverse Events by System<br>Organ Class, Preferred Term and Age Group (65<br>Years Old) | Incidence of Serious Adverse Events by System<br>Organ Class, Preferred Term and BMI |
| Table 14.3.1.3.5 | Table 14.3.1.4 | Table 14.3.1.5 | Table 14.3.1.6 | Table 14.3.1.7.1 | Table 14.3.1.7.2 | Table 14.3.1.8 | Table 14.3.1.8.1 | Table 14.3.1.8.2 | Table 14.3.1.8.3 | Table 14.3.1.8.4.1 | Table 14.3.1.8.4.2 | Table 14.3.1.8.5 |


DocuSign Envelope ID: 0709CFD0-5808-479E-B07C-DD202170566C

Protocol AVE-901-104 Phase 3 Open-Label Avenue Therapeutics, Inc.

Tramadol Infusion 07FEB2019

| Table 14.3.2.1.1 | Chemistry Laboratory Parameters: Results and Change from Baseline to End of Treatment | Safety Population | Unique |
|---|---|---|---|
| Table 14.3.2.1.2 | Shift from Baseline to End of Treatment in Serum<br>Chemistry Parameters | Safety Population | Repeat |
| Table 14.3.2.1.3 | Potentially Clinically Significant Results in<br>Chemistry values | Safety Population | Unique |
| Table 14.3.2.2.1 | Hematology Laboratory Parameters: Results and Change from Baseline to End of Treatment | Safety Population | Repeat |
| Table 14.3.2.2.2 | Shift from Baseline to End of Treatment in Hematology Parameters | Safety Population | Repeat |
| Table 14.3.2.2.3 | Potentially Clinically Significant Results in<br>Hematology values | Safety Population | Unique |
| Table 14.3.2.3.1 | Urinalysis Parameters: Continuous Results and Change from Baseline to End of Treatment | Safety Population | Repeat |
| Table 14.3.2.3.2 | Urinalysis Parameters: Categorical Results | Safety Population | Repeat |
| Table 14.3.2.3.3 | Shift from Baseline to End of Treatment in Urinalysis Parameters | Safety Population | Repeat |
| Table 14.3.2.3.4 | Potentially Clinically Significant Results in Urinalysis values | Safety Population | Unique |
| Table 14.3.3.1 | Vital Signs: Results and Change from Baseline | Safety Population | Repeat |
| Table 14.3.3.2 | Potentially Clinically Significant Results in Vital Signs | Safety Population | Unique |
| Table 14.3.4.1 | 12-Lead ECG Exam: Results and Change from Baseline | Safety Population | Repeat |
| Table 14.3.4.2 | ECG Interpretation in 12-Lead ECG Exam | Safety Population | Repeat |
| Table 14.3.4.3 | Potentially Clinically Significant Results in 12-<br>Lead ECG Exam | Safety Population | Repeat |


Tramadol Infusion 07FEB2019

# 14.1.2. Figures

| Figure NumberFigure TitleStudy PopulationFigure 14.2.1Cumulative Proportion of Subjects (%) Versus Total Exposure (mg)Safety Population | | | |
|---|---|---|---|
| tion of Subjects (%) Versus Total Exposure (my | Figure Number | Figure Title | ly Populatio |
| | Figure 14.2.1 | tion of Subjects (%) Versus Total Exposure (my | Safety Population |


Tramadol Infusion 07FEB2019

14.1.3. Listings

| Listing Number | T : | Study Population |
|---|---|---|
| | Listing 11the | |
| Listing 16.2.1 | Screening, Informed Consent and Study Population | All Screened Subjects |
| Listing 16.2.2.1 | List of Inclusion/Exclusion Eligibility Criteria | |
| Listing 16.2.2.2 | Subjects not Meeting I/E or Pre-Operative Criteria | Safety Population |
| Listing 16.2.3 | Local Laboratory Tests for Eligibility checking | Safety Population |
| Listing 16.2.4 | Protocol Deviations | Safety Population |
| Listing 16.2.5 | Subject Completion/Early Termination | Safety Population |
| Listing 16.2.6 | Demographics and Baseline Characteristics | Safety Population |
| Listing 16.2.7 | Medical/Surgical History | Safety Population |
| Listing 16.2.8 | Opioid History | Safety Population |
| Listing 16.2.9 | Pregnancy Test | Safety Population |
| Listing 16.2.10 | ASA Physical Status | Safety Population |
| Listing 16.2.11 | Surgery Information | Safety Population |
| Listing 16.2.12 | Prior and Concomitant Medications | Safety Population |
| Listing 16.2.13 | Non-Medication Therapy | Safety Population |
| Listing 16.2.14 | Study Drug Administration | Safety Population |
| Listing 16.2.15 | Summary of Study Drug Exposure | Safety Population |
| Listing 16.2.16 | Patient Global Assessment (PGA) | Safety Population |
| Listing 16.2.17 | Adverse Events | Safety Population |
| Listing 16.2.18 | Serious Adverse Events | Safety Population |
| Listing 16.2.19 | At Least Possibly Related Treatment Emergent Adverse Events | Safety Population |
| Listing 16.2.20 | Adverse Events Leading to Study Discontinuation | Safety Population |
| Listing 16.2.21 | Adverse Events Leading to Death | Safety Population |
| Listing 16.2.22 | Adverse Events Related to Local Tolerability at The Infusion Site | Safety Population |
| Listing 16.2.23.1 | Chemistry Laboratory Results | Safety Population |
| Listing 16.2.23.2 | Hematology Laboratory Results | Safety Population |
| Listing 16.2.23.3 | Urinalysis Laboratory Results | Safety Population |
| Listing 16.2.24 | Vital Signs | Safety Population |
| Listing 16.2.25 | Physical Examination | Safety Population |
| Listing 16.2.26 | 12-Lead ECG Exam Assessments | Safety Population |


Tramadol Infusion 07FEB2019

# 15. DOCUMENT HISTORY

| Version<br># | Summary of Changes | Section Changed | Date |
|--------------|--------------------|-----------------|-----------|
| 1.0 | Initial Version | NA | 07FEB2019 |




#### **Certificate Of Completion**

Envelope Id: 0709CFD05808479EB07CDD202170566C

Subject: Please DocuSign: AVE-901-104\_SAP\_Final\_v1.0\_07FEB2019.pdf

Source Envelope:

Document Pages: 43 Signatures: 6 Envelope Originator:

Certificate Pages: 5 Initials: 0 Angela Geekie

AutoNav: Enabled

Envelopeld Stamping: Enabled

Time Zone: (UTC-08:00) Pacific Time (US & Canada)

100 W California Blvd., Unit 25

Pasadena, CA 91105 ageekie@lotuscr.com IP Address: 162.236.6.81

#### **Record Tracking**

Status: Original

2/8/2019 2:15:21 PM

Holder: Angela Geekie ageekie@lotuscr.com

Location: DocuSign

Status: Completed

### **Signer Events**

Song Liou sliou@lotuscr.com

Lotus Clinical Research

Security Level: Email, Account Authentication

(Required)

Signature

Song Lion

Timestamp

Sent: 2/8/2019 2:19:55 PM Viewed: 2/8/2019 2:23:14 PM Signed: 2/8/2019 2:23:43 PM

Signature Adoption: Pre-selected Style

Signature ID:

85C80776-CFA1-404F-B9C3-4B43BB0AA100

Using IP Address: 108.51.237.84

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I am the author of this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 2/16/2018 10:40:34 AM

ID: 33003533-520a-46d0-b1ac-311cccf15c53

Jennifer Neyger

Sent: 2/8/2019 2:23:45 PM Viewed: 2/8/2019 3:42:40 PM Signed: 2/8/2019 3:43:01 PM

Jennifer Nezzer jnezzer@lotuscr.com

5:28

Lotus Clinical Research, LLC-Sub Account

Security Level: Email, Account Authentication (Required)

Signature Adoption: Pre-selected Style

Signature ID:

F51546CD-923C-410C-87CA-B1F62D450C79

Using IP Address: 45.18.125.80

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):
I have reviewed this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 8/16/2017 8:46:58 AM

ID: a2e3d9e3-0ef1-4b5e-8f0a-26d3d9799cc6

**Signer Events Signature Timestamp** Mike Ryan Sent: 2/8/2019 3:43:03 PM Mike Kyan mryan@avenuetx.com Viewed: 2/11/2019 11:58:16 AM Security Level: Email, Account Authentication Signed: 2/11/2019 11:58:46 AM (Required) Signature Adoption: Pre-selected Style Signature ID: 98E11534-E665-4F4C-B563-1912227540F0 Using IP Address: 24.60.209.159 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document **Electronic Record and Signature Disclosure:** Accepted: 11/2/2018 7:58:35 AM ID: 54379013-b0bb-49dc-9a20-08ac0d4f48b0 Scott Reines. MD Sent: 2/11/2019 11:58:49 AM Scott Reines, MD Viewed: 2/11/2019 5:34:28 PM sreines11@comcast.net Security Level: Email, Account Authentication Signed: 2/11/2019 5:36:47 PM (Required) Signature Adoption: Pre-selected Style Signature ID: A89AE03A-5748-4F3F-94C5-585073F8D59F Using IP Address: 71.224.78.90 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document **Electronic Record and Signature Disclosure:** Accepted: 9/13/2017 6:24:03 PM ID: 78ad1b50-1d57-46fa-9da1-74d2ad85eb72 Lucy Lu, MD Sent: 2/11/2019 5:36:49 PM lucy lu, MI) Viewed: 2/11/2019 6:47:45 PM llu@avenuetx.com -5DDA3F62E50E4AB. Security Level: Email, Account Authentication Signed: 2/11/2019 6:48:37 PM (Required) Signature Adoption: Pre-selected Style Signature ID: 5DDA3F62-E50E-4ABB-BCEE-9D8284AEA67B Using IP Address: 108.29.13.105 Signed using mobile With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document **Electronic Record and Signature Disclosure:** Accepted: 2/11/2019 6:47:45 PM ID: 8aa420e4-82fb-478f-b678-bbae84fb1184 Mark Harnett Sent: 2/11/2019 6:48:39 PM Mark Harriett markharnett@comcast.net Viewed: 2/12/2019 4:19:37 AM Avenue Signed: 2/12/2019 4:20:06 AM Security Level: Email, Account Authentication Signature Adoption: Pre-selected Style (Required) Signature ID: 0D9F4DA5-2C0A-4BDD-8A63-BE5F1FE45B64 Using IP Address: 73.249.51.37 With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document

| Electronic Record and Signature Disclosure:<br>Accepted: 11/22/2017 4:07:14 AM<br>ID: 8a82d85c-7ccb-45dd-a23b-b96e2e583e40 | | |
|---|---|---|
| In Person Signer Events | Signature | Timestamp |
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Notary Events | Signature | Timestamp |
| Notary Events Envelope Summary Events | Signature<br>Status | Timestamps |
| | • | · |
| Envelope Summary Events Envelope Sent Certified Delivered Signing Complete | Status Hashed/Encrypted Security Checked Security Checked | Timestamps 2/11/2019 6:48:39 PM 2/12/2019 4:19:38 AM 2/12/2019 4:20:06 AM |

Timestamp

Signature

Signer Events

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

Please read the information below carefully and thoroughly. By checking the "I agree to use Electronic Records and Signatures" box in the DocuSign system, you confirm you can access this information electronically to your satisfaction and agree to these terms and conditions below.

#### **Getting paper copies**

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after signing session. If you wish for us to send you paper copies of any such documents from our office to you, please contact your Lotus Lead Project Manager.

# Withdrawing your consent

If you decide to receive documents from us electronically, you may at any time change your mind and tell us thereafter that you want to receive documents only in paper format. If you want to withdraw your consent and receive future documents in paper format, please contact your Lotus Lead Project Manager.

# Consequences of changing your mind

If you elect to receive documents only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the documents to you in paper format, and then wait until we receive back from you and your execution of such paper documents. To indicate to us that you are changing your mind within the DocuSign system, you must withdraw your consent using the DocuSign "Withdraw Consent" form on the signing page of a DocuSign envelope instead of signing it. This will indicate to us that you have withdrawn your consent to receive documents electronically from us and you will no longer be able to use the DocuSign system to receive documents electronically from us or to sign electronically documents from us.

# All documents will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all documents that require your signature during the course of our relationship with you. All documents will be sent to you through your e-mail as recorded in the study-specific Study Contact Sheet. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

# **How to contact Lotus Clinical Research, LLC:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically:

#### To advise Lotus Clinical Research, LLC of your new e-mail address

To let us know of a change in your e-mail address, you must send an email message to your Lotus Lead Project Manager and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.

In addition, you must notify DocuSign, Inc. to arrange for your new email address to be reflected

in your DocuSign account by following the process for changing e-mail in the DocuSign system.

# To request paper copies from Lotus Clinical Research, LLC

To request delivery from us of paper copies of the documents previously provided by us to you electronically, you must send an e-mail to your Lotus Lead Project Manager and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number.

#### To withdraw your consent

To inform us that you no longer want to receive future documents in electronic format via DocuSign you may:

i. decline to sign a document from within your DocuSign session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send an email to your Lotus Lead Project Manager withdrawing consent, and in the body of such request you must state your e-mail, full name, US Postal Address, and telephone number.

Required hardware and software

| Required naturate and software | |
|---|---|
| Operating Systems: | Windows® 2000, Windows® XP, Windows |
| | Vista® Mac OS® X |
| Browsers: | Final release versions of Internet Explorer® 6.0 |
| | or above (Windows only); Mozilla Firefox 2.0 |
| | or above (Windows and Mac); Safari <sup>TM</sup> 3.0 or |
| | above (Mac only) |
| PDF Reader: | Acrobat® or similar software may be required |
| | to view and print PDF files |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | Allow per session cookies |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, you will be asked to re-accept the disclosure. Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

# Acknowledging your access and consent to receive materials electronically

By checking the "I agree to use Electronic Records and Signatures" box in the DocuSign system, you are confirming to us that:

- You can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC CONSUMER DISCLOSURES document; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify Lotus Clinical Research, LLC, as described above, you consent to receive through electronic means documents that require your signature